CLINICAL TRIAL: NCT04105842
Title: Refitting Daily Disposable Contact Lens Wearers With Dry Eye Disease With A Different Daily Disposable Lens Type
Acronym: CORGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 41251
Record Dates: First submitted 2019-09-13; First posted 2019-09-26 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Masking Description: Participants will be masked to the lens type (brand) they will be wearing during the study in order to reduce bias towards or against this product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Delfilcon A (Experimental): All study participants will be refit with Delfilcon A (Dailies Total 1) lenses which they will wear for 1 month.
  Interventions: Device: Delfilcon A

INTERVENTIONS:
Device: Delfilcon A — Participants wear delafilcon A contact lenses on a daily disposable basis.
  Other Names: Dailies Total 1

SUMMARY:
The purpose of this study is to refit habitual wearers of daily disposable contact lenses who currently experience symptoms of dry eye and discomfort during lens wear with a different type of daily disposable contact lens. Ocular signs and symptoms of dry eye will be assessed following the guidelines outlined by the Tear Film and Ocular Surface Society (TFOS) in the Dry Eye Workshop II (DEWS II). The performance of the habitual contact lenses and the study lenses will be determined using different optometric assessments. Study lenses will be worn for one month following a daily disposable wear schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. As per TFOS DEWS II, have dry eye symptoms (without CL wear) as determined by an OSDI score of ≥13 and at least one of the following:

   1. Tear osmolarity ≥ 308mOsm/L or interocular difference >8 mOsm/L
   2. Non-invasive tear breakup time of < 10 seconds in at least one eye
   3. More than 5 spots of corneal staining OR > 9 conjunctival spots in at least one eye
5. Reports dryness while wearing DD CLs with CLDEQ-8 score ≥ 12 and ≤ 203
6. Habitually wears soft spherical DD CLs with a power between +6.00D and -10.00D
7. Manifest spectacle cyl ≤1.00DC in either eye
8. BCVA ≤0.20 log MAR each eye with habitual & DT1
9. Acceptable fit with habitual & DT1
10. Willing to wear DT1 CLs at least 3 days per week and 6 hours per day throughout the study

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by self-report);
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Has taken part in another clinical research study within the last 14 days;
10. Current habitual wearer of DT1
11. Any ocular and/or systemic conditions or concomitant medication to contraindicate contact lens wear or be expected to interfere with the primary outcome variables.

    * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single site between September 2019 and June 2022. The first participant was enrolled on September 23, 2019 and the last participant was enrolled on June 23, 2022.
Pre-assignment Details: Out of 40 participants enrolled, 37 met the inclusion criteria.
Groups:
- Delefilcon A: All study participants will be refit with Delefilcon A (Dailies Total 1) lenses which they will wear for 1 month.
  Delefilcon A: Participants wear delefilcon A contact lenses on a daily disposable basis.
Period: Overall Study
Arm/Group | Delefilcon A
Started | 37
Completed | 35
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Delfilcon A
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 37

OUTCOME MEASURES:

1. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1 after screening with habitual lenses
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
score on a scale | 72.5 [20 to 90]

2. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 3 after screening with habitual lenses
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
score on a scale | 73.5 [20 to 100]

3. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 5 after screening with habitual lenses
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
score on a scale | 80 [20 to 100]

4. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: 1-week follow up with habitual lens
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
score on a scale | 75 [25 to 90]

5. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 85 [20 to 100]

6. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 3 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [35 to 100]

7. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 5 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [40 to 100]

8. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [40 to 100]

9. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 21 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [50 to 100]

10. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 28 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [30 to 100]

11. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: 1-month follow up with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [40 to 100]

12. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1 after screening with habitual lenses
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
score on a scale | 70 [10 to 90]

13. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 3 after screening with habitual lenses
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
score on a scale | 70 [20 to 100]

14. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 5 after screening with habitual lenses
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
score on a scale | 70 [25 to 100]

15. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: 1-week follow up with habitual lens
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
score on a scale | 70 [20 to 95]

16. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [30 to 100]

17. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 3 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [20 to 100]

18. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 5 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 75 [35 to 100]

19. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 70 [40 to 100]

20. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 21 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [40 to 100]

21. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 28 after dispense with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [20 to 100]

22. Primary Outcome: Subjective Rating of End of Day Dryness With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: 1-month follow up with delefilcon A
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
score on a scale | 80 [40 to 100]

23. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 1 after screening with habitual lenses
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
hours per day | 10.9 [6.0 to 18.0]

24. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 3 after screening with habitual lenses
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
hours per day | 11.4 [6.0 to 18.4]

25. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 5 after screening with habitual lenses
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
hours per day | 11.4 [6.0 to 17.5]

26. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: 1-week follow up with habitual lens
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
hours per day | 12 [3.2 to 16.5]

27. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 1 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 11.0 [6.7 to 17.4]

28. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 3 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 10.4 [5.5 to 18.1]

29. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 5 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 12.0 [6.0 to 17.5]

30. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 7 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 11.7 [6.0 to 18.0]

31. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 21 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 12.1 [6.0 to 17.3]

32. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: Day 28 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 12.0 [4.3 to 17.2]

33. Primary Outcome: Average Lens Wear Time
Description: Average lens wear time is recorded
Time Frame: 1-month follow up with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 12.5 [6.5 to 17.0]

34. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 1 after screening with habitual lenses
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
hours per day | 7.0 [1.0 to 14.6]

35. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 3 after screening with habitual lenses
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
hours per day | 6.8 [0.8 to 15.5]

36. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 5 after screening with habitual lenses
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
hours per day | 6.4 [1.3 to 15.3]

37. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: 1-week follow up with habitual lens
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 36
hours per day | 6.0 [1.0 to 12.5]

38. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 1 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 7.5 [1.2 to 15.5]

39. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 3 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 7.0 [1.2 to 18.1]

40. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 5 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 7.5 [0.8 to 17.5]

41. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 7 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 8.1 [2.3 to 16.1]

42. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 21 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 7.3 [0.9 to 16.7]

43. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: Day 28 after dispense with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 7.3 [1.0 to 17.2]

44. Primary Outcome: Comfortable Lens Wear Time
Description: Comfortable lens wear time (Time of discomfort - Time of insertion)
Time Frame: 1-month follow up with delefilcon A
Measure: Median (Full Range); unit: hours per day
Arm/Group | Delfilcon A
Number analyzed (Participants) | 35
hours per day | 8.5 [1.0 to 17.0]

ADVERSE EVENTS:
Time Frame: Up to 35-48 days
Description: Regular investigator assessment. An adverse event was defined as any unfavourable and unintended sign, symptom, or disease temporarily associated with a study procedure, whether there was a causal relationship or not.
Groups:
- Ocular Adverse Events Only: Habitual Contact Lenses; Systemic Adverse Events: Habitual Contact Lenses: All study participants will wear their habitual daily disposable contact lenses for 6-14 days.
- Ocular Adverse Events Only: Delefilcon A; Systemic Adverse Events: Delefilcon A: All study participants will be refit with Delefilcon A (Dailies Total 1) lenses which they will wear for 1 month.
  Delefilcon A: Participants wear delefilcon A contact lenses on a daily disposable basis.
Arm/Group | Ocular Adverse Events Only: Habitual Contact Lenses | Ocular Adverse Events Only: Delefilcon A | Systemic Adverse Events: Habitual Contact Lenses | Systemic Adverse Events: Delefilcon A
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35 | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35 | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 1/37 | 1/35 | 0/37 | 0/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocular Adverse Events Only: Habitual Contact Lenses (N=37) | Ocular Adverse Events Only: Delefilcon A (N=35) | Systemic Adverse Events: Habitual Contact Lenses (N=37) | Systemic Adverse Events: Delefilcon A (N=35)
Stye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Asymptomatic raised spot in left lower lid.
Foreign body trail (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Foreign body trail on cornea (epithelium).

LIMITATIONS AND CAVEATS:
The study was affected by the COVID-19 pandemic, which resulted in a mandated site closure to limit the spread of COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT04105842/Prot_SAP_000.pdf